CLINICAL TRIAL: NCT01029782
Title: Intravenous Cefazolin Plus Oral Probenecid vs. Oral Cephalexin for the Treatment of Cellulitis: a Randomized Controlled Trial
Brief Title: Comparison of Intravenous Cefazolin Plus Oral Probenecid With Oral Cephalexin for the Treatment of Cellulitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kelowna General Hospital (Other Government)
Collaborators: Canadian Society of Hospital Pharmacists (Other); Capital Health, Canada (Other); Interior Health Authority, Canada (Unknown)
Responsible Party: Principal Investigator, Dawn Dalen, Clinical Pharmacy Specialist, Emergency Medicine, Kelowna General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KGHQEII-0001
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Cellulitis
Keywords: Cellulitis; Emergency Department; Cefazolin; Probenecid; Cephalexin
MeSH Terms: conditions — Cellulitis; Emergencies | interventions — Cefazolin; Probenecid; Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV cefazolin plus oral probenecid and placebo cephalexin (Active Comparator)
  Interventions: Drug: IV cefazolin plus oral probenecid and placebo cephalexin
- Oral cephalexin and saline IV plus probenecid placebo (Active Comparator)
  Interventions: Drug: Oral cephalexin and saline IV plus probenecid placebo

INTERVENTIONS:
Drug: IV cefazolin plus oral probenecid and placebo cephalexin — Intravenous cefazolin 2 g IV plus probenecid 1 g daily plus cephalexin placebo orally four times daily.
  Arms: IV cefazolin plus oral probenecid and placebo cephalexin
Drug: Oral cephalexin and saline IV plus probenecid placebo — Cephalexin 500 mg orally four times daily plus saline IV and oral probenecid placebo daily
  Arms: Oral cephalexin and saline IV plus probenecid placebo

SUMMARY:
The purpose of this study is to determine whether oral cephalexin is equivalent to intravenous cefazolin plus oral probenecid for the treatment of uncomplicated skin and soft tissue infections in patients that present to the emergency department.

DETAILED DESCRIPTION:
Skin and soft tissue infections (SSTIs) are a common reason for presentation to an Emergency Department (ED) in Canada. Although many patients with mild SSTI are able to be managed at home with oral antibiotics, those with mild-moderate infections are often treated with parenteral antibiotics. Current practice patterns in Canadian EDs indicate this patient population is often treated with intravenous cefazolin once daily along with oral probenecid and return to the ED or other ambulatory setting for daily medication administration and assessment. This parenteral regimen has been found to result in success rates comparable to studies which have evaluated treatment success with oral antibiotics in this patient population (89-97%). Although successful outcome can be achieved with this approach, it is often inconvenient for the patient to return to the ED/ambulatory care unit daily and does contribute to overall ED/ambulatory care visit volumes and overall health care costs. Unfortunately, there has never been a study which has evaluated the relative efficacy and safety or oral antibiotics to the aforementioned parenteral approach in this patient population and thus there remains a significant knowledge gap which must be addressed before a change in current practice can be explored.

The objective of the study is to determine whether oral cephalexin is equivalent to intravenous cefazolin plus oral probenecid for the treatment of uncomplicated SSTIs in patients that present to the ED. This study will be a prospective, multi-centered, randomized controlled non-inferiority trial comparing cephalexin 500 mg orally four times to cefazolin 2 g IV plus probenecid 1 g orally, in patients presenting to the ED with presumed diagnosis of SSTI. The primary outcome will be to compare the proportion of patients failing therapy for their cellulitis after 72 hours of antibiotic treatment with oral cephalexin or IV cefazolin/oral probenecid 1 g daily. Secondary outcomes include the clinical cure rate at 7 days, percentage of patients requiring hospital admission, percentage of patients stepped down to oral antibiotics on or before day 7 of therapy, percentage of patients requiring an additional antibiotic prescription on day 7, and the frequency of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with a presumed diagnosis of mild to moderate skin and soft tissue infection
* Deemed well enough to be treated as an outpatient
* 19 years of age or older

Exclusion Criteria:

* known allergy to study drugs
* known chronic kidney disease with a creatinine clearance <30 mL/min
* known previous methicillin-resistant staphylococcus aureus (MRSA) infection
* use of antibiotics for greater than 24 hours in the past 7 days
* wound/abscess requiring operative debridement or incision and drainage
* suspected necrotizing fasciitis, osteomyelitis or septic arthritis
* febrile neutropenia
* concomitant documented bacteremia
* Two or more signs of systemic sepsis
* new altered mental status
* infections at a site involving prosthetic materials
* animal or human bite wound infections
* post-operative wound infections
* known peripheral vascular disease
* superficial thrombophlebitis
* pregnant/breastfeeding
* obesity (BMI > 30 kg/m2)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Dalen, PharmD, Principal Investigator — Interior Health; Peter Zed, PharmD, Principal Investigator — Capital Health, Canada
Locations (2):
- Canada (2):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia

REFERENCES:
- [Derived] Dalen D, Fry A, Campbell SG, Eppler J, Zed PJ. Intravenous cefazolin plus oral probenecid versus oral cephalexin for the treatment of skin and soft tissue infections: a double-blind, non-inferiority, randomised controlled trial. Emerg Med J. 2018 Aug;35(8):492-498. doi: 10.1136/emermed-2017-207420. Epub 2018 Jun 18. PMID 29914924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included if they presented to the ED with presumed diagnosis of mild-moderate SSTI and were deemed well enough to be treated as outpatients and be able to return to the ED daily.
Period: Overall Study
Arm/Group | IV Cefazolin Plus Oral Probenecid and Placebo Cephalexin | Oral Cephalexin and Saline IV Plus Probenecid Placebo
Started (All patients randomized were allocated to study arms) | 102 | 104
Completed (All patients remaining in the study arms at the 72 hour endpoint) | 99 | 96
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — Diagnosis changed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Three patients in the cephalexin arm were removed, as 2 had exclusion criteria found prior to the first doses of study medication were given and 1 patient withdrew consent in the first 24 hours.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Cefazolin Plus Oral Probenecid and Placebo Cephalexin | Oral Cephalexin and Saline IV Plus Probenecid Placebo | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.21 (17.71) | 52.01 (19.64) | 53.62 (18.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 30 | 66
  Male | 66 | 71 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 102 | 101 | 203

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Failing Therapy After 72 Hours of Antibiotic Treatment With Oral Cephalexin or Intravenous Cefazolin Plus Oral Probenecid.
Time Frame: 72 hours
Population: Per-Protocol Analysis at 72 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Cefazolin Plus Oral Probenecid and Placebo Cephalexin | Oral Cephalexin and Saline IV Plus Probenecid Placebo
Number analyzed (Participants) | 99 | 96
Participants | 6 | 4

ADVERSE EVENTS:
Arm/Group | IV Cefazolin Plus Oral Probenecid and Placebo Cephalexin | Oral Cephalexin and Saline IV Plus Probenecid Placebo
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/101
Other Adverse Events (participants affected / at risk) | 4/102 | 5/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Cefazolin Plus Oral Probenecid and Placebo Cephalexin (N=102) | Oral Cephalexin and Saline IV Plus Probenecid Placebo (N=101)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomit (Gastrointestinal disorders) | 3 (3) | 1 (1)
Infusion Reaction (Vascular disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No